CLINICAL TRIAL: NCT01135823
Title: Symptom Assessment With Patient Surveys
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Christina Baggott NP RN, Stanford University School of Medicine
Other Study IDs: SU-07292009-3461; 97085; PEDSVAR0001
Record Dates: First submitted 2010-06-01; First posted 2010-06-03 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-06

CONDITIONS: Carcinomas; Squamous Cell Carcinoma; Adenocarcinoma
MeSH Terms: conditions — Carcinoma; Carcinoma, Squamous Cell; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Patient survey

SUMMARY:
The primary purpose of the proposed research is to explore methods of obtaining symptom assessments from pediatric oncology patients and/or their caregivers in hopes of improving the accuracy and thoroughness of these reports. Additionally the researchers hope to simply staff efforts in obtaining detailed medical histories from pediatric oncology patients.

ELIGIBILITY:
Inclusion Criteria:

* Approximately 150 patients ages 0-18 years (75 for each group-intervention and control) will be enrolled.
* These patients will be pediatric oncology patients who have received chemotherapy within the prior four weeks and being seen in the oncology clinic for an out-patient visit.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: These patients will be pediatric oncology patients who have received chemotherapy within the prior four weeks and being seen in the oncology clinic for an out-patient visit.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Baggott NP RN, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States